CLINICAL TRIAL: NCT02117544
Title: Evaluation of Visual Performance With a Multifocal High ADD Soft Contact Lens Design
Brief Title: Multifocal High ADD Contact Lens Proof of Concept Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C-13-057
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Presbyopia
Keywords: Contact lens; Presbyopia; Multifocal
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- New MF, then AOAMF (Other): Lotrafilcon B multifocal contact lenses (new), followed by lotrafilcon B multifocal contact lenses. Each product worn bilaterally (in both eyes) for about 1 hour.
  Interventions: Device: Lotrafilcon B multifocal contact lenses (new); Device: Lotrafilcon B multifocal contact lenses
- AOAMF, then New MF (Other): Lotrafilcon B multifocal contact lenses, followed by lotrafilcon B multifocal contact lenses (new). Each product worn bilaterally (in both eyes) for about 1 hour.
  Interventions: Device: Lotrafilcon B multifocal contact lenses (new); Device: Lotrafilcon B multifocal contact lenses

INTERVENTIONS:
Device: Lotrafilcon B multifocal contact lenses (new)
Device: Lotrafilcon B multifocal contact lenses
  Other Names: AIR OPTIX® AQUA Multifocal; AOAMF

SUMMARY:
The purpose of this study is to evaluate the visual performance of a new multifocal High ADD contact lens compared to the currently-marketed AIR OPTIX® AQUA MULTIFOCAL (AOAMF) High ADD Contact Lens.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent document;
* Presbyopic and require at least 2.25 diopters (D) spectacle ADD power;
* Current or previous soft contact lens wearer;
* Not able to achieve monocular near visual acuity (VA) 0.2 logarithm of the Minimum Angle of Resolution (logMAR) [Early Treatment of Diabetic Retinopathy Study (ETDRS)] or better in each eye with AIR OPTIX® AQUA Multifocal (AOAMF) High ADD Contact Lenses;
* Willing and able to wear multifocal contact lenses in both eyes within the available range of powers for this trial;
* Manifest cylinder less than or equal to 1.00 D;
* Able to achieve best corrected visual acuity (BCVA) of 20/25 or better in each eye at distance (as determined by manifest refraction);
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, disease, or abnormality that contraindicates contact lens wear within 6 months prior to enrollment, as determined by the investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator; or any use of topical ocular medications that would require instillation during contact lens wear;
* Any history of herpetic keratitis;
* History of corneal or refractive surgery, irregular cornea or unilateral pseudophakia;
* Biomicroscopy findings (except for corneal vascularization) that are moderate (Grade 3) or severe (Grade 4);
* Corneal vascularization that is mild (Grade 2) or higher;
* A pathologically dry eye that precludes contact lens wear;
* Monocular (only 1 eye with functional vision);
* Anisometropia ≥ 1.50 D (contact lens distance prescription);
* Clinically significant (> 1 millimeter) anisocoria;
* History of intolerance or hypersensitivity to any component of the investigational products;
* Concurrent participation in a contact lens or contact lens care product clinical trial within the previous 30 days;
* Eye injury or ocular or intra-ocular surgery within 6 months prior to enrollment;
* Any ocular or systemic medical condition that may, in the opinion of the Investigator, preclude safe administration of the study lenses or affect the results of this study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, Vision Care, GCRA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 7 study centers located in the US.
Pre-assignment Details: Of the 268 enrolled, 159 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (109).
Groups:
- New MF, Then AOAMF: Lotrafilcon B multifocal contact lenses (new), followed by lotrafilcon B multifocal contact lenses. Each product worn bilaterally for about 1 hour.
- AOAMF, Then New MF: Lotrafilcon B multifocal contact lenses, followed by lotrafilcon B multifocal contact lenses (new). Each product worn bilaterally for about 1 hour.
Period: Period 1
Arm/Group | New MF, Then AOAMF | AOAMF, Then New MF
Started | 54 | 55
Treated | 52 | 55
Completed | 52 | 55
Not Completed | 2 | 0
Not completed — Lost to follow-up (prior to treatment) | 2 | 0
Period: Period 2
Arm/Group | New MF, Then AOAMF | AOAMF, Then New MF
Started | 52 | 55
Completed | 52 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and treated subjects.
Groups:
- Overall: AIR OPTIX® AQUA Multifocal and lotrafilcon B Multifocal (new design) contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: High Contrast Visual Acuity (HCVA) Near Monocular
Description: Visual Acuity (clarity or sharpness of vision) was measured at high contrast level. HCVA was assessed monocularly (each eye separately) at 40 centimeters using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart and measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value indicates better visual acuity. Both eyes contributed to the analysis.
Time Frame: Day 1, 10 minutes after lens insertion, each product
Population: This analysis population includes all randomized subjects excluding those who met the critical deviation criteria as specified in the Deviations and Evaluability Plan (DEP).
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- New MF: Lotrafilcon B multifocal (new design) contact lenses worn during Period 1 or Period 2 for 1 hour
- AOAMF: Lotrafilcon B multifocal contact lenses worn during Period 1 or Period 2 for 1 hour
Arm/Group | New MF | AOAMF
Number analyzed (Participants) | 104 | 104
Number analyzed (Eyes) | 208 | 208
logMAR | 0.18 (0.02) | 0.32 (0.02)

2. Secondary Outcome: HCVA Distance Monocular
Description: Visual Acuity (clarity or sharpness of vision) was measured at high contrast level. HCVA was assessed monocularly (each eye separately) at 6 meters using an ETDRS chart and measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value indicates better visual acuity. Both eyes contributed to the analysis.
Time Frame: Day 1, 10 minutes after lens insertion, each product
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | New MF | AOAMF
Number analyzed (Participants) | 104 | 104
Number analyzed (Eyes) | 208 | 208
logMAR | 0.11 (0.01) | 0.06 (0.01)

3. Secondary Outcome: HCVA Intermediate Monocular
Description: Visual Acuity (clarity or sharpness of vision) was measured at high contrast level. HCVA was assessed monocularly (each eye separately) at 1 meter using an ETDRS chart and measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value indicates better visual acuity. Both eyes contributed to the analysis.
Time Frame: Day 1, 10 minutes after lens insertion, each product
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | New MF | AOAMF
Number analyzed (Participants) | 104 | 104
Number analyzed (Eyes) | 208 | 208
logMAR | 0.04 (0.01) | 0.02 (0.01)

4. Secondary Outcome: Low Contrast Visual Acuity (LCVA) Distance Monocular
Description: Visual Acuity (clarity or sharpness of vision) was measured at low contrast level. LCVA was assessed monocularly (each eye separately) at 6 meters using an ETDRS chart and measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value indicates better visual acuity. Both eyes contributed to the analysis.
Time Frame: Day 1, 10 minutes after lens insertion, each product
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | New MF | AOAMF
Number analyzed (Participants) | 104 | 104
Number analyzed (Eyes) | 208 | 208
logMAR | 0.44 (0.01) | 0.39 (0.01)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (3 months). AEs are reported as pre-treatment and treatment-emergent, based on treatment-specific exposure.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained as solicited comments from subjects and as observations by the study Investigator as outlined in the study protocol.
Groups:
- Pre-treatment: Includes all enrolled subjects/eyes prior to exposure to the investigational products
- New MF: Includes all subjects/eyes exposed to New MF
- AOAMF: Includes all subjects/eyes exposed to AOAMF
Arm/Group | Pre-treatment | New MF | AOAMF
Serious Adverse Events (participants affected / at risk) | 0/268 | 0/107 | 0/107
Other Adverse Events (participants affected / at risk) | 0/268 | 0/107 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.